CLINICAL TRIAL: NCT01805349
Title: Study of the Association Between Digital Osteoarthritis and Lower Limb Osteoarthritis (Knee and Hip) in Terms of Severity and Evolution - Khoala Group Ancillary Project / Cohort Khoala
Brief Title: Study of Association Between Digital Osteoarthritis and Lower Limb Osteoarthritis
Acronym: Khoala
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-AOI-01
Record Dates: First submitted 2013-02-28; First posted 2013-03-06 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Digital Arthrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- X-Rays (Other): patients with digital arthrosis and hip/knee arthrosis will practice hand X-rays
  Interventions: Radiation: Hand X-rays

INTERVENTIONS:
Radiation: Hand X-rays — Hand X-rays to assess the digital arthrosis

SUMMARY:
Among the risk factors for lower limb osteoarthritis, if obesity is probably the most studied, digital osteoarthritis received increasing interest in recent years. Recent publications have highlighted a link between obesity and digital osteoarthritis, but also a very probable link between digital osteoarthritis and structural progression of knee osteoarthritis. Few data including hip exist and need to be confirmed on larger scale studies. We have with "Khoala" a national multiregional cohort of symptomatic gonarthrosis and coxarthrosis representative of the general population (which is rarely the case in the literature) including X ray, clinical and biological follow-up (hips and / or knees).

ELIGIBILITY:
Inclusion Criteria:

* men or women aged 40 to 75 years
* with symptomatic osteoarthritis of the hip and / or knee (femoro-tibial), unilateral or bilateral
* with a confirmed diagnosis (criteria of the American College of Rheumatology :ACR) and Kellgren and Lawrence radiological stage ≥ 2.

Exclusion Criteria:

* painful hip or knee prosthesis
* osteotomy in the past

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2013-11-04 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2013-12-01 (Actual)

PRIMARY OUTCOMES:
Kellgren and Lawrence score | Change at 2 years
  Kellgren and Lawrence score for hip or knee

SECONDARY OUTCOMES:
Harris score | Harris score at 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of rheumatology, nice university hospital, Nice, France